CLINICAL TRIAL: NCT03641300
Title: Cognitive Outcomes and Response/Remission Efficacy of Convulsive Therapies for Bipolar Depression: the CORRECT-BD Trial
Brief Title: Efficacy of Convulsive Therapies for Bipolar Depression
Acronym: CORRECT-BD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University of British Columbia (Other); Ontario Shores Centre for Mental Health Sciences (Other); Brain Canada (Other)
Responsible Party: Principal Investigator, Daniel Blumberger, Medical Head and Co-Director, Temerty Centre for Therapeutic Brain Intervention, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 015-2018
Record Dates: First submitted 2018-08-17; First posted 2018-08-22 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Bipolar Disorder; Bipolar Depression; Bipolar I Disorder; Bipolar II Disorder
Keywords: Magnetic Seizure Therapy; Electroconvulsive Therapy; Bipolar Disorder; Depression; Suicidal Ideation
MeSH Terms: conditions — Bipolar Disorder; Depression; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: The study is a randomized, double blind, parallel-group clinical trial with two treatment arms conducted at three academic institutions: the Temerty Centre for Therapeutic Brain Intervention based at CAMH in Toronto, ON; the Ontario Shores Centre for Mental Health Sciences in Whitby, Ontario; and UBC Hospital based at the University of British Columbia in Vancouver, BC. CAMH aims to recruit 40 participants. Parkwood Institute and UBC Hospital aim to recruit 30 participants each.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will be randomized into the study using a permuted block method with a random number generator. The study statistician will prepare the randomization scheme. The block size will be fixed and study personnel will be blinded to the randomization block size
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Magnetic Seizure Therapy (MST) (Experimental): MST treatments will be administered using the MagPro MST with Cool TwinCoil.
  Interventions: Device: Magnetic Seizure Therapy (MST)
- Electroconvulsive Therapy (ECT) (Active Comparator): ECT treatments will be administered using the MECTA spECTrum 5000Q or MECTA Sigma
  Interventions: Device: Electroconvulsive Therapy (ECT)

INTERVENTIONS:
Device: Magnetic Seizure Therapy (MST) — MST treatment will be administered using the MagPro MST with a Cool TwinCoil over the frontal cortex in the midline position using 100 Hz stimulation. The MST determination of seizure threshold will be done using 100% machine output applied at 100 Hz at progressively escalating train durations, commencing at 2 seconds and increasing by 2 seconds with each subsequent stimulation until an adequate seizure is produced. During subsequent sessions, one stimulation will be delivered using a train duration that is 4 seconds longer than the train duration at threshold (with a maximum train duration of 10 seconds).
  This will be performed under the effect of anesthesia. The treatment procedure is approximately 10 minutes, followed by a recovery period of approximately 30 minutes.
  Other Names: MST
  Arms: Magnetic Seizure Therapy (MST)
Device: Electroconvulsive Therapy (ECT) — In the ECT arm treatment, the MECTA spectrum 5000Q machine will be used, which is an FDA approved device used for providing standard-of-care clinical ECT treatments. The ECT determination of seizure threshold and the adjustment of energy at subsequent sessions will be based on a standard published protocol. All participants will receive RUL-UB ECT at six times the seizure threshold under the effect of anesthesia. The treatment procedure is approximately 10 minutes, followed by a recovery period of approximately 30 minutes
  Other Names: ECT
  Arms: Electroconvulsive Therapy (ECT)

SUMMARY:
This trial aims to assess the efficacy and tolerability of Magnetic Seizure Therapy (MST) as an alternative to electroconvulsive therapy (ECT) for Bipolar Disorder (BD). Research indicates that the prevalence of treatment resistance in bipolar depression is twice that of unipolar depression. The limited effectiveness of current treatments for bipolar depression coupled with the medical and economic burden associated with the disorder engenders a need for novel therapeutic interventions that can provide greater response and remission rates.

DETAILED DESCRIPTION:
The study will involve a randomized, double blind, non-inferiority clinical trial with two treatment arms conducted in three academic institutions (the Centre for Addiction and Mental Health (CAMH) in Toronto, Ontario; the Ontario Shores Centre for Mental Health Sciences in Whitby, Ontario; and University of British Columbia (UBC) Hospital in Vancouver, British Columbia). The investigators are pursuing a non-inferiority clinical trial in an effort to compare MST to right unilateral ultrabrief pulse ECT (RUL-UB-ECT). Treatment will be administered two to three days per week. Depression symptoms will be assessed with the 24-item Hamilton Depression Rating Scale (HRSD-24) and suicidality will be assessed with the Scale for Suicidal Ideation (SSI). Remission will be defined as HRSD-24 < or = 10 and a > 60% decrease in scores from baseline on two consecutive ratings. Once a participant reaches remission, a second rating to confirm remission will be conducted immediately before their next scheduled treatment. If remission is confirmed, they will then be considered a completer of the acute treatment course. Remission of suicidal ideation is defined as a score of 0 on the SSI. Therefore, there will be no specific minimum number of treatments that patients must receive to be classified as remitters. However, patients who do not meet remission criteria after 21 treatment sessions will be considered non-remitters and will cease treatment sessions. This maximum treatment number was chosen allowing for the possibility that MST may require more treatment sessions to achieve remission, similar to RUL-UB ECT. The blind will not be broken to participants until the completion of the entire study.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included if they:

1. are inpatients or outpatients;
2. are voluntary and competent to consent to treatment and research procedures according to ECT/MST attending psychiatrist;
3. have a MINI International Neuropsychiatric Interview diagnosis, Version 6 (MINI-6.0) diagnosis of non-psychotic Bipolar Disorder (Type I or II)
4. are 18 years of age or older
5. have a baseline HRSD-24 score > 21;
6. are considered to be appropriate to receive convulsive therapy as assessed by an ECT attending psychiatrist and a consultant anaesthesiologist
7. are agreeable to keeping their current antidepressant treatment constant during the intervention;
8. are likely able to adhere to the intervention schedule;
9. meet the MST safety criteria;
10. If a woman of child-bearing potential: is willing to provide a negative pregnancy test and agrees not to become pregnant during trial participation.

Exclusion Criteria:

Patients will be excluded if they:

1. have a history of MINI diagnosis of substance dependence or abuse within the past three months;
2. have a concomitant major unstable medical illness;
3. are pregnant or intend to get pregnant during the study;
4. have a MINI diagnosis of any primary psychotic disorder
5. have a MINI diagnosis of obsessive compulsive disorder, or post-traumatic stress disorder deemed to be primary and causing more functional impairment than the depressive disorder
6. have probable dementia based on study investigator assessment;
7. have any significant neurological disorder or condition likely to be associated with increased intracranial pressure or a space occupying brain lesion, e.g., cerebral aneurysm;
8. present with a medical condition, a medication, or a laboratory abnormality that could cause a major depressive episode or significant cognitive impairment in the opinion of the investigator (e.g., hypothyroidism with low TSH, rheumatoid arthritis requiring high dose prednisone, or Cushing's disease);
9. have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed;
10. require a benzodiazepine with a dose greater than lorazepam 2 mg/day (or equivalent benzodiazepine) or any anticonvulsant due to the potential of these medications to limit the efficacy of both MST and ECT;
11. are unable to communicate in English fluently enough to complete the neuropsychological tests;
12. have a non-correctable clinically significant sensory impairment (i.e., cannot hear or see well enough to complete the neuropsychological tests).

    These eligibility criteria are congruent with the criteria that have been used in the major ECT trials conducted during the past decade;
13. elevated mood, defined as a score of 20 or higher on the Young Mania Rating Scale (YMRS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
Remission (score </= 10) on the Hamilton Rating Scale for Depression - 24 (HRSD-24) | Greater than 8 treatments (2.5 weeks)
  Hamilton Rating Scale for Depression (24-item version):
  * This scale is used to quantify the severity of symptoms of depression
  * Scale range: 0-76 (total score)
  * Lower scores indicate lower severity of depressive symptoms (i.e., better outcome)
  * Higher scores indicate higher severity of depressive symptoms (i.e., worse outcome)
Cognitive adverse effects as indexed by the Autobiographical Memory Test (AMT) | Greater than 8 treatments (2.5 weeks)
  Autobiographical Memory Test:
  - Interviewer-rated measure with 10 items that indexes autobiographical memory recall and specificity.

SECONDARY OUTCOMES:
Improvement in symptom severity of Suicidal Ideation as measured by the Scale for Suicidal Ideation (SSI) | 7 weeks
  Scale for Suicidal Ideation:
  * This scale is used to assess the presence or absence of suicidal ideation and the degree of severity of suicidal ideas
  * Scale range: 0 - 38 (total score)
  * Lower scores indicate lower severity of suicidal ideation (i.e., better outcome)
  * Higher scores indicate higher severity of suicidal ideation (i.e., worse outcome)
Number of self-reported and clinical-reported adverse events | Up to 7 weeks
  Number of adverse events in both treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Blumberger, MD, MSc, Principal Investigator — Centre for Addiction and Mental Health
Locations (3):
- Canada (3):
  - UBC Hospital, University of British Columbia (UBC), Vancouver, British Columbia
  - Temerty Centre for Therapeutic Brain Intervention, Centre for Addiction and Mental Health, Toronto, Ontario
  - Ontario Shores Centre for Mental Health Sciences, Whitby, Ontario

REFERENCES:
- [Derived] Jiang J, Zhang C, Li C, Chen Z, Cao X, Wang H, Li W, Wang J. Magnetic seizure therapy for treatment-resistant depression. Cochrane Database Syst Rev. 2021 Jun 16;6(6):CD013528. doi: 10.1002/14651858.CD013528.pub2. PMID 34131914
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital — http://www.camh.net/research